CLINICAL TRIAL: NCT02730325
Title: A Randomized, Double-Blind, Placebo-Controlled Study to Evaluate the Impact of Serum-derived Bovine Immunoglobulin/Protein Isolate (SBI) on Clostridium Difficile (C. Difficile) Infection (CDI) in Hospitalized Ulcerative Colitis (UC) Patients
Brief Title: To Evaluate the Impact of SBI on C. Difficile in Hospitalized UC Patients
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Study terminated due to limited enrollment.
Sponsor: Northwestern University (Other)
Collaborators: Entera Health, Inc (Industry)
Responsible Party: Principal Investigator, Stephen Hanauer, Professor of Medicine, Northwestern University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: STU00200335
Record Dates: First submitted 2016-02-05; First posted 2016-04-06 (Estimated); Last update posted 2021-11-18 (Actual); Status verified 2021-11

CONDITIONS: Clostridium Difficile
Keywords: CDI; C. diff; Ulcerative Colitis; UC; IBD; Inflammatory Bowel Disease
MeSH Terms: conditions — Colitis, Ulcerative; Inflammatory Bowel Diseases

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- SBI 10 g BID (Active Comparator): Serum-derived bovine immunoglobulin/protein isolate (SBI) 10.0 grams twice per day
  Interventions: Other: Serum-derived bovine immunoglobulin/protein isolate (SBI)
- Placebo BID (Placebo Comparator): Placebo
  Interventions: Other: Placebo

INTERVENTIONS:
Other: Serum-derived bovine immunoglobulin/protein isolate (SBI)
  Arms: SBI 10 g BID
Other: Placebo
  Arms: Placebo BID

SUMMARY:
The effects of serum-derived bovine immunoglobulin/protein isolate (SBI) will be evaluated and compared to matching placebo in two distinct patient populations:

I. Hospitalized ulcerative colitis (UC) patients who tested positive for Clostridium difficile (C. difficile) at time of admission and are receiving vancomycin.

II. Hospitalized UC patients who tested negative for C. difficile at time of admission.

DETAILED DESCRIPTION:
The effects of serum-derived bovine immunoglobulin/protein isolate (SBI) will be evaluated and compared to matching placebo in two distinct patient populations:

I. Hospitalized ulcerative colitis (UC) patients who tested positive for Clostridium difficile (C. difficile) at time of admission and are receiving vancomycin.

Primary Objective:

• To evaluate the effect of SBI on time (# of days) to resolution of diarrhea, defined as a consecutive 24 hour period with only formed bowel movements (Bristol Stool Scale (BSS) ≤ 4) in this patient population

Secondary Objectives:

* To evaluate the ability of SBI to decrease the incidence of recurrent C. difficile infection (CDI) following successful treatment with vancomycin.
* To evaluate the effect of SBI on UC status
* To evaluate the effect of SBI on nutritional status
* To evaluate the safety and tolerability of SBI
* To evaluate the effect of SBI on subjects' quality of life (QOL)
* To investigate the effect of SBI in fecal microbiome
* To evaluate the length of hospitalization (time of hospitalization to time of discharge)

II. Hospitalized UC patients who tested negative for C. difficile at time of admission.

Primary Objective:

• To evaluate the effect of SBI on time (# of days) to resolution of diarrhea, defined as a consecutive 24 hour period with only formed bowel movements (Bristol Stool Scale (BSS) ≤ 4) in this patient population

Secondary Objectives:

* To evaluate the effect of SBI in decreasing the incidence of CDI
* To evaluate the effect of SBI on UC status
* To evaluate the effect of SBI on nutritional status
* To evaluate the safety and tolerability of SBI
* To evaluate the effect of SBI on subjects' QOL
* To investigate the effect of SBI in fecal microbiome
* To evaluate the length of hospitalization (time of hospitalization to time of discharge)

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of UC confirmed by colonoscopy and histology.
* Confirmed active UC upon hospital admission, defined by a partial Mayo Score of ≥ 3 with a stool frequency subscore of ≥ 2.
* Concomitant therapy for UC will be permitted. Subjects will be instructed not to make any medication changes after hospital discharge before first discussing with the Investigator.
* Eligible subjects will be assigned to one of two different and independent patient groups based on C. difficile status as determined by clinical symptoms with diarrhea and laboratory tests: either a polymerase chain reaction (PCR) assay or glutamate dehydrogenase (GDH) screening test used in two- or three-step algorithm with subsequent toxin A and B EIA testing.

Exclusion Criteria:

* Subjects with history of constipation within a week of the screening visit; or any serious hepatic, renal, cardiovascular, neurological or hematological disorder in the opinion of the Investigator.
* Subjects with history of drug or alcohol abuse, history of psychiatric disorders, known allergy or hypersensitivity to beef or any component of SBI.
* Subjects with a history of antibiotic treatment within the 4 weeks prior to enrollment.
* Subjects using anti-diarrheal medications (e.g., loperamide and bismuth subsalicylate).

  * Note: anti-diarrheal medications will be prohibited throughout the study.
* Subjects who have been admitted to the hospital more than 48 hours prior to enrollment.
* Women who are pregnant.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2015-12 (Actual); Primary Completion 2017-12-12 (Actual); Study Completion 2018-01-05 (Actual)

PRIMARY OUTCOMES:
Time (# of days) to resolution of diarrhea | 12 weeks
  Group 1 & Group 2 subjects: Stool consistency will be assessed using the BSS. Subjects will be provided a daily diary A to record the time and consistency of each bowel movement in a 24 hour period. At the Week 4 visit, the Investigator will calculate the time (# of days) to resolution of diarrhea, defined as a consecutive 24 hour period with only formed bowel movements (BSS ≤ 4), after initiation of investigational product (Day 1).

SECONDARY OUTCOMES:
Incidence of recurrent CDI | 12 weeks
  Group I subjects: if subject develops diarrhea (≥ 3 unformed stools in 24h period) at any point following successful treatment with vancomycin. The presence of C. difficile will be determined by PCR or GDH/Toxin EIA.
Incidence of C. difficile | 12 weeks
  Group II subjects: Incidence of C. difficile will be determined following 12 weeks of investigational product. Symptoms will be assessed by daily diary and by P SCCAI at each study visit. Should the subject develop diarrhea (≥ 3 unformed stools in 24h period) at any point during the study participation, he/she will return to the clinic and be tested for C. difficile by PCR or GDH/Toxin EIA.
UC status measured by P-SCCAI | 4, 8 and 12 weeks
  Group I & Group II subjects
UC status measured by BSS | 4 weeks
  Group I & Group II subjects
UC status measured by Fecal calprotectin | 12 weeks
  Group I & Group II subjects
UC status measured by CRP | 12 weeks
  Group I & Group II subjects
UC status measured by colectomy rate | 12 weeks
  Group I & Group II subjects
Nutritional Status measured by pre-albumin | 12 weeks
  Group I & Group II subjects
Nutritional Status measured by albumin | 12 weeks
  Group I & Group II subjects
Nutritional Status measured by hand grip strength | 12 weeks
  Group I & Group II subjects
Nutritional Status measured by fecal alpha-1 antitrypsin | 12 weeks
  Group I & Group II subjects
Safety and Tolerability evaluated by reported and observed treatment related adverse events | 12 weeks
  Group I & Group II subjects
Quality of Life evaluated using the SF-36 | 12 weeks
  Group I & Group II subjects
Fecal Microbiome | 12 weeks
  Group I & Group II subjects
Length of Hospitalization | 12 weeks
  Group I & Group II subjects

CONTACTS AND LOCATIONS:
Overall Officials: Stephen B Hanauer, MD, Principal Investigator — Northwestern University
Locations (3):
- United States (3):
  - University of Miami, Miami, Florida
  - Northwestern University, Chicago, Illinois
  - Rush University, Chicago, Illinois